CLINICAL TRIAL: NCT03193827
Title: In-line Filtration Reduces Postoperative Venous Peripheral Phlebitis Associated With Cannulation: a Randomised Clinical Trial
Brief Title: In-line Filtration Reduces Postoperative Phlebitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Careggi Hospital (Other)
Responsible Party: Principal Investigator, Gianluca Villa, MD, Careggi Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEAV IN17/0000015
Record Dates: First submitted 2017-06-18; First posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Phlebitis
Keywords: vip score; peripheral venous cannulation; particles
MeSH Terms: conditions — Phlebitis

STUDY DESIGN:
Intervention Model Description: Two hundred and sixty-eight patients undergoing surgery are randomised 1:1 to in-line filtration (study group) and standard care (control group). For patients randomize to in-line filtration, in-line filters (Pall, Dreieich, Germany) are used during anaesthesia and the following 96 postoperative hours. Patients randomize to standard care (control group) are managed without an in-line filter and according to local routine practice for intravenous drug administration in the adult patient. The incidence and severity of phlebitis are evaluated using the Visual Infusion Phlebitis (VIP) Score23 every 12 hrs from the end of surgery until 96 hrs postoperatively in both groups. Time and severity of phlebitis and time and causes for venous cannula removal are all compared between groups.
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): In this group in-line filters (Pall, Dreieich, Germany) are connected to peripheral vascular access and used during anaesthesia and the following 96 postoperative hours.
  Interventions: Device: In-line filtration
- control group (Active Comparator): Patients randomised to standard care are managed without an in-line filter and according to local routine practice for intravenous drug administration in the adult patient.
  Interventions: Device: Standard treatment

INTERVENTIONS:
Device: In-line filtration — In-line filtration is used during anesthesia and postoperative 96 hrs in study group to purify endovascular fluids administrations reducing postoperative phlebitis
  Arms: study group
Device: Standard treatment — Patients are treated with standard intravenous solutions and vascular access management
  Arms: control group

SUMMARY:
The aim of this study is to demonstrate the efficacy of in-line filtration in reducing the incidence of postoperative phlebitis associated with peripheral short-term vascular access.

In this controlled trial, 268 surgical patients are 1:1 randomised to in-line filtration (study group) and standard care (control group). The incidence of phlebitis (defined as Visual Infusion Phlebitis, VIP score≥2) within 48hrs postoperatively is compared between the two groups, as well as the onset and severity of phlebitis and the reasons for removal of the cannula. The lifespan of venous cannulae and cost-of-care are compared for the study and control groups through a Kaplan-Meier curve. Multivariate Cox regression analysis is performed to evaluate the effect of in-line filtration on risk of phlebitis and cannula removal.

DETAILED DESCRIPTION:
A randomised, controlled, clinical trial is performed at the Department of Anesthesia and Intensive Care of the Azienda Ospedaliero-Universitaria Careggi in Florence, Italy, to assess the effects of in-line filtration on the incidence of postoperative phlebitis. The Ethical Committee of the institution has approved the study (CEAV IN17/0000015). Patients preoperatively sign consent forms for participation in this trial.

An incidence of phlebitis equal to 50% within 48 hrs from peripheral venous cannulation has been preliminarily described in our centre during standard care (unpublished data). Two hundred and sixty-eight patients undergoing surgery are 1:1 randomised to in-line filtration (study group) and standard care (control group) to observe a 20% reduction in postoperative phlebitis within 48 hrs after surgery in the study group through a one-side chi-square analysis with statistical power of 90% and statistical significance of 0.025.

Every surgical patient scheduled for surgery, who preoperatively signed the consent form and underwent peripheral venous cannulation, is considered for this study. Patients undergoing central venous catheterisation or long-/middle-term peripheral cannulation are excluded.

On the day of surgery, all enrolled patients undergo standard peripheral venous cannulation according to the up-to-date standard of care. After placement of venous cannula and before the induction of anaesthesia, patients are randomised for in-line filtration or standard care.

For patients randomized to in-line filtration, in-line filters (Pall, Dreieich, Germany) are used during anaesthesia and the following 96 postoperative hours.

Patients randomised to standard care (control group) are managed without an in-line filter and according to local routine practice for intravenous drug administration in the adult patient. The enrolment in this study don't influence the type of anaesthesia or the postoperative pharmacological treatment previously scheduled for the patient.

The incidence and severity of phlebitis are evaluated using the Visual Infusion Phlebitis (VIP) Score every 12 hrs from the end of surgery until 96 hrs postoperatively. The postoperative VIP score evaluations are performed by another author, blinded to each patient's randomisation group. This filter are held by containment bands on the patient's arm and are completely covered by a breathable dressing medication to maintain the evaluator blind on the patient's randomisation group. The dressing medication never covers the vein where the cannulae are placed. Transparent dressing is used for cannula medication to allow cannulation site inspection

Phlebitis is defined as a VIP score ≥2. The primary end-point of the study is to assess the incidence of phlebitis in the 48 postoperative hours using a Fisher's exact test. Time and severity of phlebitis and time and causes for venous cannula removal are all compared between groups. In particular, data distribution is assessed through the Shapiro-Wilk test. Continuous data are presented as a median and interquartile range (IQR) or mean ± standard deviation (SD) and analysed through a Mann-Whitney or Student's t-test, according to data distribution. Qualitative data are presented as percentages and analysed through chi-square analysis. The Bonferroni adjustment is used for multiple comparisons. The lifespan of the cannulae is described for the study and the control groups through the Kaplan-Meier curve. Multivariate Cox regression analysis with a backwards selection is performed to evaluate the effect of in-line filtration on the risk of phlebitis and cannula removal, independently from other factors. Results are presented as p-value, hazard ratio (HR) and 95% confident interval (95%CI)

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old
* Consent to trial participation and randomization obtained in preoperative period

Exclusion Criteria:

* Pregnancy
* Presence of central vascular access with central or peripheral iserction
* Presence of long peripheral vascular access such as Midline or MiniMidline
* Patients envolved in other comparative trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-10 (Actual)

PRIMARY OUTCOMES:
The aim of the trial is to demonstrate the efficacy of in-line filtration in reducing the incidence of postoperative phlebitis associated with peripheral short-term vascular access in the 48 postoperative hours | VIP score is evaluated every 12hrs from the end of surgery until 96 hrs postoperatively
  The incidence of phlebitis is evaluated through Visual Infusion Phlebitis (VIP) score.Phlebitis is defined as a VIP score ≥ 2. A Fischer's exact test will be use to evaluate difference between study group and control group.

SECONDARY OUTCOMES:
A secondary objective is to evaluate difference between study group and control group phlebitis onset in the 96 postoperative hours | VIP score is evaluated every 12hrs from the end of surgery until 96 hrs postoperatively
  The incidence of phlebitis is evaluated through Visual Infusion Phlebitis (VIP) score.Phlebitis is defined as a VIP score ≥ 2. A Fischer's exact test will be use to evaluate difference between study group and control group.
A secondary objective is to show difference between study group and control group phlebitis severity in the 96 postoperative hours | VIP score is evaluated every 12hrs from the end of surgery until 96 hrs postoperatively
  The incidence of phlebitis is evaluated through Visual Infusion Phlebitis (VIP) score.Phlebitis is defined as a VIP score ≥ 2. A Fischer's exact test will be use to evaluate difference between study group and control group.
A secondary objective is to evaluate care cost increase secondary to in-line filtration management between study group and control group | In 96 postoperative hours, all materials used (infusion sets, vascular dressing devices, filters, kit for venipuncture...) to manage vascular access in control group and in study group is registered
  Care cost is calculated through evaluation of intravenous treatment expenditure in control group and study group. In both group is calculated the costs of the disposables used and the costs of the time spent by the staff involved in the management of peripheral venous access during the first 96 hours postoperatively. In these evaluation we consider: frequency of infusion set substitutions and all devices used; frequency of vascular access replacement, alla devices used to replace a new cannulae and caregiver cost related to time needed to replacement and cost for hours of nursing, medical or anesthesiological work.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Niel-Weise BS, Stijnen T, van den Broek PJ. Should in-line filters be used in peripheral intravenous catheters to prevent infusion-related phlebitis? A systematic review of randomized controlled trials. Anesth Analg. 2010 Jun 1;110(6):1624-9. doi: 10.1213/ANE.0b013e3181da8342. Epub 2010 Apr 30. PMID 20435946
- [Derived] Villa G, Chelazzi C, Giua R, Tofani L, Zagli G, Boninsegni P, Pinelli F, De Gaudio AR, Romagnoli S. In-Line Filtration Reduces Postoperative Venous Peripheral Phlebitis Associated With Cannulation: A Randomized Clinical Trial. Anesth Analg. 2018 Dec;127(6):1367-1374. doi: 10.1213/ANE.0000000000003393. PMID 29697508